CLINICAL TRIAL: NCT01631617
Title: Effects of Treatments on the Microbiome in Healthy Volunteers and Patients With Atopic Dermatitis
Brief Title: Effects of Treatments on Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120159; 12-AR-0159
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-30

CONDITIONS: Eczema; Dermatitis; Skin Diseases, Genetic; Dermatitis, Atopic; Skin Diseases
Keywords: Investigator-Blinded; Skin Biopsy; Randomized; Antibiotics; Topical
MeSH Terms: conditions — Eczema; Dermatitis; Skin Diseases, Genetic; Dermatitis, Atopic; Skin Diseases | interventions — Trimethoprim; Sulfamethoxazole; Cephalexin; Doxycycline; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 1A/Cephalexin (Active Comparator): Cephalexin + Placebo bleach
  Interventions: Drug: Cephalexin
- 1B/TMP/SMX (Active Comparator): TMP/SMZ DS 800 /160 orally every 12 hours for 14 days
  Interventions: Drug: Trimethoprim/sulfamethoxazole (TMP/SMZ)
- 1C/Doxycycline 100 (Active Comparator): Doxycycline 100 mg orally every 12 hours for 56 days
  Interventions: Drug: Cephalexin; Other: Sodium hypochlorite
- 1D/Doxycycline 20 (Active Comparator): Doxycycline 20 mg orally every 12 hours for 56 days
  Interventions: Drug: Doxycycline
- 2A/Cephalexin + Dilute bleach (Active Comparator): Systemic antibiotics (Cephalexin) + dilute bleach study bath liquid
  Interventions: Drug: Cephalexin; Other: Sodium hypochlorite
- 2B/Cephalexin + Placebo bleach (Placebo Comparator): Systemic antibiotics (Cephalexin) + placebo study bath liquid
  Interventions: Drug: Cephalexin; Other: Placebo Sodium hypochlorite
- 2C/Placebo capsules + Dilute bleach (Placebo Comparator): Placebo capsules + dilute bleach study bath liquid
  Interventions: Other: Sodium hypochlorite; Other: Placebo capsules
- 2D/Placebo capsules + Placebo bleach (Placebo Comparator): Placebo capsules + placebo study bath liquid
  Interventions: Other: Placebo capsules; Other: Placebo Sodium hypochlorite
- 3A/Cephalexin + Dilute bleach (Active Comparator): Systemic antibiotics (Cephalexin) + dilute bleach study bath liquid
  Interventions: Drug: Cephalexin; Other: Sodium hypochlorite
- 3B/Cephalexin + Placebo bleach (Placebo Comparator): Systemic antibiotics (Cephalexin) + placebo study bath liquid
  Interventions: Drug: Cephalexin; Other: Placebo Sodium hypochlorite

INTERVENTIONS:
Drug: Trimethoprim/sulfamethoxazole (TMP/SMZ) — 800/160 orally every 12 hours for 14 days
  Arms: 1B/TMP/SMX
Drug: Cephalexin — 500 mg orally every 8 hours for 14 days
  Arms: 1A/Cephalexin; 1C/Doxycycline 100; 2A/Cephalexin + Dilute bleach; 2B/Cephalexin + Placebo bleach; 3A/Cephalexin + Dilute bleach; 3B/Cephalexin + Placebo bleach
Drug: Doxycycline — 20 mg orally every 12 hours for 56 days or 100 mg orally every 12 hours for 56 days
  Arms: 1D/Doxycycline 20
Other: Sodium hypochlorite — 6 % dilute bleach
  Arms: 1C/Doxycycline 100; 2A/Cephalexin + Dilute bleach; 2C/Placebo capsules + Dilute bleach; 3A/Cephalexin + Dilute bleach
Other: Placebo capsules — Capsule orally every 8 hours daily for 14 days
  Arms: 2C/Placebo capsules + Dilute bleach; 2D/Placebo capsules + Placebo bleach
Other: Placebo Sodium hypochlorite — Three times a week for 14 days
  Arms: 2B/Cephalexin + Placebo bleach; 2D/Placebo capsules + Placebo bleach; 3B/Cephalexin + Placebo bleach

SUMMARY:
Background:

- Atopic dermatitis, or eczema, is a chronic skin disorder. Patients sometimes have infections with S. aureus bacteria. Researchers want to study how eczema treatments affect the number and the type of bacteria on the skin.

Objectives:

- To study the effect of eczema treatments on skin bacteria.

Eligibility:

* Individuals between 2 and 25 years of age who have moderate to severe atopic dermatitis.
* Healthy volunteers between 18 and 40 years of age with no history of eczema.

Design:

* Participants will be screened with a physical exam and medical history. Research samples will be collected. Skin biopsies may also be performed.
* All participants will be assigned to one of several study groups.
* Healthy volunteers must not have taken antibiotics in the year before the start of the study.
* All participants will have regular study visits during their 1-year participation. More research samples will be collected at these visits.
* Healthy volunteers may be asked to come in for a one-time follow up after the 1 year mark.

DETAILED DESCRIPTION:
BACKGROUND:

* The use of antibiotics has revolutionized medicine, yet the impact of antimicrobials on the human microbiome is incompletely understood.
* Antimicrobial treatments, including topical and systemic antibiotics, are highly effective and are frequently used to manage disease flares of atopic dermatitis (AD). Concomitant use of dilute bleach baths reduces the clinical severity of AD in patients with clinical signs of bacterial skin infections.
* The longitudinal impact of various antimicrobials on the human microbiome, particularly in skin, has not been systematically investigated.
* Our recent study demonstrated that antibiotic-resistant bacteria can be observed after antibiotic exposure; however, multi-year persistence has not been evaluated

OBJECTIVES:

Primary:

- To characterize microbiome alterations in healthy adult volunteers and patients with AD after antimicrobial treatments.

ELIGIBILITY:

* All subjects must be co-enrolled in NIH protocol 08-HG-0059
* (Cohorts 1 [NO FURTHER ACCRUAL], 2 [INACTIVE], 4 [NO FURTHER ACCRUAL], 5 [INACTIVE]) Healthy volunteers aged 18 to 50 years with no history of AD.
* (Cohort 1 [NO FURTHER ACCRUAL], 2 [INACTIVE], 4 [NO FURTHER ACCRUAL] and 5 [INACTIVE]) No prior use of systemic antibiotics in preceding 12 months.
* (Cohort 3 [INACTIVE]) Subjects 2-50 years with atopic dermatitis with symptoms of active bacterial infection.
* (Cohort 3 [INACTIVE]) Objective SCORAD (SCORing Atopic Dermatitis) score of >= 15 indicating moderate-to-severe disease.
* (Cohort 6) Individuals previously enrolled in Cohorts 1 [NO FURTHER ACCRUAL] and 4 [NO FURTHER ACCRUAL].

DESIGN:

* A prospective, interventional, longitudinal study examining changes in microbiome resulting from randomized, placebo-controlled, investigator-blinded antimicrobial treatments.
* Subjects in Cohort 1 [NO FURTHER ACCRUAL] will be randomized to take one of 4 open label antibiotic regimens.
* Subjects from Cohort 2 [INACTIVE] randomized to one of four possible blinded treatment combinations of study baths and antibiotics.
* Subjects in Cohort 3 [INACTIVE] will be randomized to a cephalexin regimen with or without study baths.
* Subjects in Cohorts 4 [NO FURTHER ACCRUAL] and 5 [INACTIVE] will receive one of two open label antibiotic regimens.
* All subjects will undergo longitudinal microbiome sampling.
* Subjects who completed on-protocol antibiotic regimen in Cohorts 1 [NO FURTHER ACCRUAL] and 4 [NO FURTHER ACCRUAL] may be recruited >1 year after completion of Cohorts 1 and 4 to undergo an optional single visit for microbiome sampling as Cohort 6.
* AD patients [INACTIVE] will undergo clinical assessment to determine responses of skin infections to treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cohorts 1 [NO FURTHER ACCRUAL], 2 [INACTIVE], 4 [NO FURTHER ACCRUAL] and 5 [INACTIVE]: Healthy Volunteers

* Males and females aged 18-50 years at time of initial protocol sampling
* Subjects must participate fully and be willing to comply with the procedures of the protocol
* Subjects must be co-enrolled in NIH protocol 08-HG-0059
* Ability of subject to understand and provide written informed consent
* Access to bathing facilities (Cohort 2 [INACTIVE])
* Ability to swallow capsules or tablets

Cohort 3 [INACTIVE]: Atopic Dermatitis Patients

* Subjects must be aged 2-50 years
* Subjects must be co-enrolled in NIH protocol 08-HG-0059
* Subjects must have a diagnosis of atopic dermatitis on the basis of the criteria defined by UK Working Party s Diagnostic Criteria for Atopic Dermatitis
* Subjects must have a primary care provider
* Subjects must have an Objective SCORAD (SCORing Atopic Dermatitis) of greater than or equal to 15 indicating AD severity of moderate to severe
* Prior to initiation of randomized treatment, subjects must have signs of bacterial skin infections (skin weeping, crusting, and/or pustules)
* Access to bathing facilities
* All subjects and/or their Legally Authorized Representative (LAR) must have the ability and agree to participate fully and comply with

the procedures of the protocol and provide informed consent. Pediatric patients will be included in age appropriate discussions and

age appropriate assent will be obtained in accordance with NIH guidelines.

-Ability of subject to understand and provide written informed consent

Cohort 6: Healthy Volunteers

* Subjects previously enrolled in Cohorts 1 [NO FURTHER ACCRUAL] and 4 [INACTIVE] who completed on-protocol antibiotic regimen
* Subjects must participate fully and be willing to comply with the procedures of the protocol
* Ability of subject to understand and provide written informed consent

EXCLUSION CRITERIA:

Cohorts 1 [NO FURTHER ACCRUAL] and 2 [INACTIVE]: Healthy Volunteers

* Does not meet inclusion criteria
* Any female with symptoms and/or serum hormone levels consistent with perimenopause or menopause
* Use of systemic antibiotics in 12 months preceding baseline sampling
* Use of swimming pools, hot tubs, or whirlpools in 7 days preceding baseline sampling
* Use of topical or oral complementary/alternative medicine (CAM) agents within 4 weeks of initiation of treatment
* Known allergic reaction to sulfa, beta-lactam, or tetracycline class drugs; or lidocaine or epinephrine
* Family history of toxic epidermal necrolysis
* Known allergy or sensitivity to sodium hypochlorite (NaOCl)
* History of AD or asthma
* Inability to comply with the requirements of the protocol
* Pregnant or lactating
* Subjects with a primary or acquired immunodeficiency, including HIV seropositiviy
* Any chronic past or present medical illness, including chronic skin diseases like psoriasis
* Subjects receiving or planning to receive an IND agent, ultraviolet light therapy, monoclonal antibodies, or systemic immunosuppressants
* Subjects who provide direct healthcare or reside in healthcare facilities or in non-hospital settings such as, assisted living facilities, homeless shelters, jails and prisons as well as subjects with frequent exposure to laboratory animals

Cohort 3 [INACTIVE]: Atopic Dermatitis Patients

* Does not meet inclusion criteria
* Any female with symptoms and/or serum hormone levels consistent with perimenopause or menopause
* Known allergic reaction to beta-lactam class drugs, lidocaine, or epinephrine
* Family history of toxic epidermal necrolysis
* Known allergic reaction to sodium hypochlorite (NaOCl)
* Use of systemic antibiotics within 8 weeks, or topical antibiotics on intended sampling sites within 3 weeks, prior to baseline sampling
* Use of topical corticosteroids on all intended sampling sites within 7 days, prior to baseline sampling
* Use of topical or oral CAM agents within 4 weeks of initiation of treatment
* Subjects with known primary or acquired immunodeficiency
* Subjects with unstable or uncontrolled medical conditions that could require hospitalization during the initial month of the study or who have been hospitalized for treatment of these conditions in the one month prior to baseline sampling
* Subjects receiving or planning to receive an IND agent, ultraviolet light therapy, monoclonal antibodies, or systemic immunosuppressants within 7 days or 5 half-lives (whichever is the longer time period) of initiating treatment on this protocol
* Subjects who are currently receiving or have received chemotherapy or radiation for treatment of malignancies within the previous 6 months
* Pregnancy or lactating

Cohorts 4 [NO FURTHER ACCRUAL] and 5 [INACTIVE]: Healthy Volunteers

* Does not meet inclusion criteria
* Any female with symptoms and/or serum hormone levels consistent with perimenopause or menopause
* Use of systemic antibiotics in 12 months preceding baseline sampling
* Use of swimming pools, hot tubs, or whirlpools in 7 days preceding baseline sampling
* Use of topical or oral complementary/alternative medicine (CAM) agents within 4 weeks of initiation of treatment
* (Cohort 4 [NO FURTHER ACCRUAL]) Known allergic reaction to sulfa class drugs; or lidocaine or epinephrine
* (Cohort 5 [INACTIVE]) Known allergic reaction to tetracycline class drugs; or lidocaine or epinephrine
* Family history of toxic epidermal necrolysis
* History of AD or asthma
* Inability to comply with the requirements of the protocol
* Pregnant or lactating
* Subjects with a primary or acquired immunodeficiency, including HIV seropositivity
* Any chronic past or present medical illness, including chronic skin diseases like psoriasis
* Subjects receiving or planning to receive an IND agent, ultraviolet light therapy, monoclonal antibodies, or systemic immunosuppressants
* Subjects who provide direct healthcare or reside in healthcare facilities or in non-hospital settings such as assisted living facilities, homeless shelters, jails and prisons as well as subjects with frequent exposure to laboratory animals

Cohort 6: Healthy Volunteers

* Does not meet inclusion criteria
* Use of swimming pools, hot tubs, or whirlpools in 7 days preceding sampling
* Use of topical or oral CAM agents within 1 week or 4 weeks, respectively, prior to sampling
* Pregnant or lactating females in all cohorts are excluded from participating due to the potential effects of the above listed antimicrobials on the developing human fetus or nursing infant; listed in Sections 11.1 through 11.5. Females of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Lactating mothers will discontinue breastfeeding prior to study enrollment.
* Smokers and subjects who use smokeless tobacco products are excluded in all cohorts due to tobacco s unknown impact on human oral mucosa and microflora.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-09-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Characterize microbiome alterations | 2 weeks
  Difference in Shannon Diversity Indices (SDI) from baseline to day 14.

SECONDARY OUTCOMES:
To obtain samples from healthy adult volunteers to evaluate and refine genomic analysis of human microbes. | Throughout the duration of the study
To examine how different antimicrobials may alter the human microbiome. | Throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Heidi H Kong, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-AR-0159.html